CLINICAL TRIAL: NCT03179748
Title: Non-interventional, Multi-Centre, Post-Authorisation Safety Study With Novoeight®/NovoEight® (Turoctocog Alfa) in Mexican Haemophilia A Patients
Brief Title: Study Investigating Novoeight®/NovoEight® (Turoctocog Alfa) in Mexican Haemophilia A Patients
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN7008-4253; U1111-1171-9845 (Other: World Health Organization (WHO))
Record Dates: First submitted 2017-05-24; First posted 2017-06-07 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Congenital Bleeding Disorder; Haemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — recombinant factor VIII N8

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- turoctocog alfa: Patients with haemophilia A
  Interventions: Drug: turoctocog alfa

INTERVENTIONS:
Drug: turoctocog alfa — Patients will be treated with commercially available turoctocog alfa according to local clinical practice at the discretion of the physician

SUMMARY:
The trial is conducted in North America. The aim of the trial is to assess the safety of turoctocog alfa under conditions of routine clinical care in patients with haemophilia A in Mexico

ELIGIBILITY:
Inclusion Criteria:

* Signed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol)
* Male and female patients with haemophilia A
* Age range is 0 years and above
* The decision to initiate treatment with commercially available turoctocog alfa has been made by the patient/Legally Acceptable Representative (LAR) and the treating physician before and independently from the decision to include the patient in this study

Exclusion Criteria:

* Previous participation in this study. Participation is defined as having given informed consent in this study
* Known or suspected allergy to turoctocog alfa or related products
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population are haemophilia A patients who based on the indication will benefit from treatment with turoctocog alfa. No limitation has been set to the severity of haemophilia A, gender, age, previously treated and untreated patients.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2021-06-16 (Actual); Study Completion 2021-06-16 (Actual)

PRIMARY OUTCOMES:
Frequency of adverse reactions | 3-36 months after enrollment
  Count and % of events

SECONDARY OUTCOMES:
Frequency of adverse events | 3-36 months after enrollment
  Count and % of events
Efficacy in treatment of bleeds | 3-36 months after enrollment
  Rated: Excellent, Good, Moderate or none
Consumption of turoctocog alfa for prophylaxis | 3-36 months after enrollment
  Measured in IU/kg/dose
Consumption of turoctocog alfa for treatment of bleeds | 3-36 months after enrollment
  Measured in IU/kg/bleeding episode
Consumption of turoctocog alfa for surgery and post-surgical period | 3-36 months after enrollment
  Measured in IU/kg
Number of patients with confirmed inhibitors | 3-36 months after enrollment
  Count of presence of inhibitors
Number of patients with allergic/hypersensitivity reactions to turoctocog alfa | 3-36 months after enrollment
  Count of episodes
Number of bleeding episodes | 3-36 months after enrollment
  Count of episodes

CONTACTS AND LOCATIONS:
Locations (1):
- Novo Nordisk Investigational Site, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com